CLINICAL TRIAL: NCT06136273
Title: Penetrating Trauma Registry and Open Source Data
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 106.TRA.2022.D
Record Dates: First submitted 2023-10-18; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Penetrating Trauma Registry and Open Source Data
Keywords: Trauma
MeSH Terms: conditions — Wounds and Injuries | interventions — Methods

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Treatment measures and intervention strategies — To conduct observational process improvement and hypothesis-deriving studies related to penetrating traumatic injuries using data from the Methodist trauma registry and open source data repositories.
  Other Names: Injury prevention

SUMMARY:
Penetrating injuries comprise roughly 30% of Methodist Health System (MHS) trauma patients. Firearm-related events have become more prevalent in the past few years. Active shooter events, mass casualties, assaults, and homicide are more commonplace which leads to an increase of trauma patients needing management of penetrating injuries.

DETAILED DESCRIPTION:
Penetrating injuries comprise roughly 30% of Methodist Health System (MHS) trauma patients. Firearm-related events have become more prevalent in the past few years . Active shooter events, mass casualties, assaults, and homicide are more commonplace which leads to an increase of trauma patients needing management of penetrating injuries. On average, penetrating traumas only make up 14% of comparable center patient volumes. In spring 2022, we also were ranked 3/10 for our penetrating trauma outcomes with lower than expected mortality (TQIP Benchmarking Report). Together, as a Level 1 trauma center with above average penetrating injury volume we must take efforts to best understand the opportunities for our patients and disseminate those observations to the trauma community

ELIGIBILITY:
Inclusion Criteria:

* • Aged 16 years or older (National Trauma Data Standard for adult)

  * Penetrating injury or intent to cause penetrating injury

Exclusion Criteria:

* • Aged 15 years or younger

  * Prisoners, pregnant persons, or other protected population
  * Not involved in penetrating trauma

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Methodist Health System (MHS) trauma patients
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-08-15 (Actual); Primary Completion 2025-08-19 (Estimated); Study Completion 2025-08-19 (Estimated)

PRIMARY OUTCOMES:
comprehensive data series | 3 years
  To establish a comprehensive data series from observational data to gain a better understanding of the specifics surrounding penetrating trauma and related events
observational process improvement | 3 years
  To conduct observational process improvement and hypothesis-deriving studies related to penetrating traumatic injuries using data from the Methodist trauma registry and open source data repositories.

CONTACTS AND LOCATIONS:
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Study data or any protected health information will not be shared with anyone that is not delegated to the study. The PI is committed to disseminate research results in a timely fashion. Sharing of results generated by the data analysis during the course of the project will be through presentation at national scientific meetings and/or publication in open access journals. All information obtained will be source de-identified and presented on a large scale and not traceable to any one particular individual.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: 2 years

REFERENCES:
- [Background] Bjelopera, J. (2022). Public Mass Shootings in the United States: Selected Implications for Federal Public Health and Safety Policy. Retrieved 18 August 2022, from https://crsreports.congress.gov/product/pdf/R/R43004.
- [Background] Lin PI, Fei L, Barzman D, Hossain M. What have we learned from the time trend of mass shootings in the U.S.? PLoS One. 2018 Oct 18;13(10):e0204722. doi: 10.1371/journal.pone.0204722. eCollection 2018. PMID 30335790
- [Background] 3. Luca, M., Malhotra, D., & Poliquin, C. (2020). The impact of mass shootings on gun policy. Journal Of Public Economics, 181, 104083. https://doi.org/10.1016/j.jpubeco.2019.104083
- [Background] AJPH Global News. Am J Public Health. 2020 Oct;110(10):1446. doi: 10.2105/AJPH.2020.305872. No abstract available. PMID 32903069
- [Background] 5. Schildkraut, J., Elsass, H., & Meredith, K. (2017). Mass shootings and the media: why all events are not created equal. Journal Of Crime And Justice, 41(3), 223-243. https://doi.org/10.1080/0735648x.2017.1284689
- [Background] Shultz JM, Thoresen S, Flynn BW, Muschert GW, Shaw JA, Espinel Z, Walter FG, Gaither JB, Garcia-Barcena Y, O'Keefe K, Cohen AM. Multiple vantage points on the mental health effects of mass shootings. Curr Psychiatry Rep. 2014 Sep;16(9):469. doi: 10.1007/s11920-014-0469-5. PMID 25085235
- [Background] 7. Silva, J. (2020). A Comparative Analysis of Foiled and Completed Mass Shootings. American Journal Of Criminal Justice, 46(2), 187-208. https://doi.org/10.1007/s12103-020-09552-2